CLINICAL TRIAL: NCT06051630
Title: Effects of Perioperative Administration of Intravenous Lidocaine in Children Operated on for Acute Generalized Peritonitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université NAZI BONI (Other)
Responsible Party: Principal Investigator, Ismael Guibla, Principal investigator, Clinical doctor, Université NAZI BONI
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INSSA 3
Record Dates: First submitted 2023-08-21; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain
Keywords: Peritonitis; Postoperative pain; Lidocaine; Burkina Faso
MeSH Terms: conditions — Pain, Postoperative; Peritonitis

STUDY DESIGN:
Intervention Model Description: This will be a randomized, double-blind clinical trial conducted at University hospital Charles De Gaulle of Ouagadougou, comparing the results of intravenous administration of lidocaine perioperatively versus administration of saline
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): The group will receive 1.5 mg/kg lidocaine 2% bolus, followed by a continuous electric syringe dose of 1.5 mg/kg/hour intraoperatively, then 1.5 mg/kg/hour during the first 24 hours postoperatively
  Interventions: Drug: Lidocaine intravenous
- Saline group (Placebo Comparator): The control group will receive an equivalent volume of saline: the volume of saline to be administered will be obtained by considering the dose of lidocaine 2% that the patient would have received if he/she had been in the interventional group.
  Interventions: Drug: Serum saline intravenous

INTERVENTIONS:
Drug: Lidocaine intravenous — Perioperative lidocaine intravenous administration
  Arms: Lidocaine group
Drug: Serum saline intravenous — Perioperative serum saline intravenous administration
  Arms: Saline group

SUMMARY:
Intravenous administration of lidocaine perioperatively after laparotomy for peritonitis could be an interesting alternative by reducing the duration of postoperative ileus, the intensity of pain and the patient's hospital stay, as well as the cost of management in our context of lack of financial, technical and human resources, hence the present study.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 6 to 15, Classified according to the American Society of Anaesthesiologists (ASA) (I, II and III) admitted for peritonitis and whose parents have given informed consent

Exclusion Criteria:

* State of shock
* Severe renal insufficiency (creatinine clearance less than 30 ml/min)
* History of allergy to lidocaine
* Refusal to participate in the study

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Resumption of transit | Up to 7 days during the postoperative period. From the date of randomization to the first postoperative gas and/or the presence of postoperative bowel sounds in the patient
  time to first gas and/or presence of bowel sounds

SECONDARY OUTCOMES:
Analog visual scale | Postoperative pain scores at 24 hours
  Average pain score, minimal value is 0, maximal value is 10 and higher score mean worse
Concentration of C-reactive protein | Hours 24 postoperative
  Average of C-reactive protein
Hospitalisation | Up to 30 days during the postoperative period. From the date of randomization to the patient's discharge from hospital or date of death
  Number of days in hospital
Postoperative mortality | Up to 30 days during the postoperative period. From date of randomization to date of death
  Number of postoperative deaths

CONTACTS AND LOCATIONS:
Overall Officials: Nazinigouba OUEDRAOGO, Professor, Study Director — JOSEPH KI-ZERBO University

IPD SHARING:
Plan to Share IPD: No